CLINICAL TRIAL: NCT04411732
Title: Myotonia, Muscle Stiffness and Elasticity in Neuromuscular Disorders
Brief Title: Myotonia and Muscle Stiffness in NMD
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Benedikt Schoser, Prof. Dr. med. Benedikt Schoser, LMU Klinikum
Other Study IDs: Version: 1 [01-JUL-2019]
Record Dates: First submitted 2020-05-25; First posted 2020-06-02 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Neuromuscular Disorders
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Walk Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with neuromuscular disorder: cohort of patients with neuromuscular disorder
  Interventions: Device: MyotonPro; Diagnostic Test: Six-minute walk test; Diagnostic Test: Semiquantitative muscle ultrasound; Diagnostic Test: Hand-held Dynamometry of muscle strength
- healthy controls: cohort of healthy controls
  Interventions: Device: MyotonPro; Diagnostic Test: Six-minute walk test; Diagnostic Test: Semiquantitative muscle ultrasound; Diagnostic Test: Hand-held Dynamometry of muscle strength

INTERVENTIONS:
Device: MyotonPro — Measurement of relaxation time, stiffness and elasticity of the following muscles, using the MyotonPro® device: on both sides thenar and hypothenar, m. biceps brachii, m. triceps brachii, m. deltoideus, m. quadriceps femoris, m. tibialis anterior and gastrocnemius muscles.
Diagnostic Test: Six-minute walk test — The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. The 6MWT has been used with a variety of other conditions than the chronic obstructive pulmonary disease (COPD) such as heart failure and stroke and is widely used in neuromuscular diseases. The six-minute-walk-test will be conducted as recommended by the American Thoracic Society. In this study, the six-minute-walk test will be performed once on visit 1 to detect the impact of muscle weakness, muscle stiffness and myotonia on muscular endurance.
Diagnostic Test: Semiquantitative muscle ultrasound — Muscle ultrasound is an ideal imaging modality that allows for atraumatic, noninvasive, radiation-free point-of-care neuromuscular imaging. Muscular dystrophies are typically associated with an increase in the echogenicity from the muscle substance, distal attenuation of muscle echo and a corresponding loss of bone echo. Spinal muscular atrophies and neuropathies also showed an increase in muscle echo along with atrophy of the muscle and increase in depth of subcutaneous tissue, but a persisting bone echo. In several other myopathies, similar changes are seen. In semi-quantitative muscle ultrasound, muscle intensity will be documented using the 4-point Heckmatt score. In addition to that, cutis, subcutaneus fat and muscle will be measured in mm.
Diagnostic Test: Hand-held Dynamometry of muscle strength — Muscle strength will be assessed by handheld dynamometry using the MicroFET2 myometer, produced by Hoggan Health Industries. This test is widely used in patients with neuromuscular diseases. To perform a test, the examiner holds the dynamometer stationary while the patient exerts a maximal force against the dynamometer. The patient makes a gradual increase in force and then completes an isometric hold for 4-5 seconds. The following muscle groups will be tested: Arm abduction, elbow flexion, elbow extension, knee extension, knee flexion, foot extension, foot flexion.

SUMMARY:
The primary objective of this study is to assess stiffness, muscle tone, relaxation periods and elasticity of various muscles in patients with dystrophic or non-dystrophic myotonia. The secondary objectives are (1) to provide reference values for stiffness, muscle tone, relaxation periods and elasticity of various muscles in patients with dystrophic or non-dystrophic myotonia; to provide reference values for stiffness, muscle tone, relaxation periods and elasticity of various muscles in patients with non-myotonic neuromuscular disorders, (3) assess correlations between to compare result values for stiffness, muscle tone, relaxation periods and elasticity with clinical muscle function tests, measured by clinical evaluation (MRC-scale) and the 6-minute walk test; (4) assess correlations between subcutaneous fat and muscle thickness and echogenicity, measured by muscle ultrasound and result values for stiffness, muscle tone, relaxation periods and elasticity.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* ≥18 years of age
* Confirmed neuromuscular disease
* written consent
* able and willing to perform study prodcedures

For healthy volunteers:

* age ≥18 years of age
* written informed consent
* no clinical sign for neuromuscular disorders

Exclusion Criteria:

* Severe comorbidities
* Patient is participating in another clinical study using investigational treatment
* Patient cannot perform required muscle function tests
* the patient, in the opinion of the investigator, is unable to adhere to the requirements of the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Approximately 70 patients will be enrolled, about 3-5 each in the following disease groups: Limb-Girdle-Muscular Dystrophy (LGMD), Myotonic Dystrophies Type 1 and 2 (DM1, DM2), Late-Onset-Pompe Disease (LOPD), Distal Myopathies, Congenital Myotonia, Spinal muscular atrophy Type 3 (SMA3), Amyotrophic lateral sclerosis (ALS) and peripheral Polyneuropathies (CIDP, HMSN). 20 healthy age- and gender-matched patients will be enrolled as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
MyotonPro device in patients with dystrophic and non-dystrophic myotonia | 1 day
  The primary objective of this study is the comparison of viscoelastic stiffness of the underlying tissue measured by stiffness (S), elasticity (D) and relaxation (R) between patients with dystrophic and non-dystrophic myotonia.

SECONDARY OUTCOMES:
MyotonPro device - reference values in patients with dystrophic and non-dystrophic myotonia | 1 day
  The secondary objective of this study is to provide reference values for stiffness, muscle tone, relaxation periods and elasticity of various muscles in patients with dystrophic or non-dystrophic myotonia.
MyotonPro device - reference values in patients with non-myotonic neuromuscular disorders | 1 day
  The secondary objective of this study is to provide reference values for stiffness, muscle tone, relaxation periods and elasticity of various muscles in patients with non-myotonic neuromuscular disorders.
MyotonPro device - correlations between stiffness, muscle tone, relaxation periods and elasticity with clinical muscle function tests | 1 day
  The secondary objective of this study is to compare stiffness, muscle tone, relaxation periods and elasticity with clinical muscle function tests, measured by clinical evaluation (MRC-scale).
MyotonPro device - correlations between stiffness, muscle tone, relaxation periods and elasticity with subcutaneous fat and muscle thickness and echogenicity | 1 day
  The secondary objective of this study is to assess correlations between subcutaneous fat and muscle thickness and echogenicity, measured by muscle ultrasound and result values for stiffness, muscle tone, relaxation periods and elasticity.
MyotonPro device - correlations between stiffness, muscle tone, relaxation periods and elasticity and the 6-minute-walk test | 1 day
  The secondary objective of this study is to compare stiffness, muscle tone, relaxation periods and elasticity with clinical muscle endurance function tests, measured by the 6-minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wenninger, Dr. med., Principal Investigator — Neurologist
Locations (1):
- Friedrich-Baur-Institute, Dep. of Neurology Klinikum der Universitaet Muenchen, Munich, Bavaria, Germany

DOCUMENTS (1):
  • Study Protocol (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT04411732/Prot_000.pdf